CLINICAL TRIAL: NCT05874973
Title: Effects of Time-controlled Adaptive Ventilation (TCAV) and Volume Control Ventilation (VCV) on the Distribution of Aerated Lung Parenchyma in Patients With Acute Respiratory Distress Syndrome (ARDS): a Pilot Study
Brief Title: Effects of TCAV and Volume Control Ventilation on the Distribution of Aerated Lung Parenchyma in ARDS Patients
Acronym: TCAV-CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, PEQUIGNOT Benjamin, Dr, Central Hospital, Nancy, France
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021PI212
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: ARDS
Keywords: Mechanical Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-Controlled Adaptative Ventilation (TCAV) (Experimental): APRV mode set with:
  * a Phigh at Plateau Pressure of the VCV mode
  * a Tlow set to terminate the expiration at 75% of the maximal expiratory flow
  * a Plow set at 0 cmH2O.
  * a Thigh set to achieve adequate decarboxylation.
  Interventions: Other: Time-controlled adaptative ventilation (TCAV)
- Volume Control Ventilation (VCV) (Active Comparator): Ventilation with the VCV mode set with:
  * a tidal volume (VT) at or below 6 ml/kg of predicted body weight
  * a positive end-expiratory pressure (PEEP) set at least at 5 cmH2O
  * a driving pressure lower than 15 cmH2O.
  Interventions: Other: Volume-controlled ventilation (VCV)

INTERVENTIONS:
Other: Time-controlled adaptative ventilation (TCAV) — Ventilation with TCAV set on the APRV mode on the ventilator.
  Arms: Time-Controlled Adaptative Ventilation (TCAV)
Other: Volume-controlled ventilation (VCV) — Ventilation with the VCV mode set on the ventilator.
  Arms: Volume Control Ventilation (VCV)

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a severe form of acute respiratory failure with mortality rates reaching as high as 35%. Management of ARDS is based on the treatment (if possible) of the underlying cause of ARDS and on invasive mechanical ventilation with positive expiratory pressure (PEEP). Another strategy of invasive ventilation, Time-Controlled Adaptative Ventilation (TCAV), is the application of specific settings to the airway pressure release ventilation (APRV) mode.

TCAV is based on a prolonged time at plateau pressure, creating a phase of continuous positive pressure, associated with brief release phases allowing the elimination of carbon dioxide. In prospective and retrospective clinical reviews, as well as in experimental animal studies, TCAV has demonstrated improvements in oxygenation and lung function, with the ability to prevent ARDS.

The thoracic computed tomography (CT) scan evaluates lung recruitment (re-aeration by positive pressure of non-ventilated lung territories) and the adverse effects of positive pressure on the parenchyma (hyperinflation).

The objective of this study is to evaluate, with CT scans performed to assess lungs of patients with ARDS, the effects of TCAV compared to a standard volumetric controlled ventilation, by measuring alveolar recruitment and over-distension.

ELIGIBILITY:
Inclusion Criteria:

* ARDS according to the Berlin definition
* invasive ventilation for no longer than 72 hours
* patient requiring a diagnostic thoracic CT scan
* consent of a family member or the person of trust
* social security affiliation

Exclusion Criteria:

* Use of iodinated contrast media injection before CT acquisitions
* ARDS criteria present during 72 hours or more
* Severe COPD
* Pneumothorax or other barotrauma-related complication
* Right ventricular failure other than acute cor pulmonale
* Absence of sedative agents and neuromuscular blockade
* Severe hemodynamic instability (norepinephrine > 0.5 µg/kg/min)
* VA-ECMO assistance
* Pregnancy
* Absence of the capacity to give consent before admission to the ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of end-expiratory non aerated lung parenchyma | during procedure (10 minutes)
  Percentage of non aerated lung parenchyma defined as % of lung at -100 to +100 Hounsfield Units (HU) divided by total lung weight, at the end of expiration.

SECONDARY OUTCOMES:
End-inspiratory overdistention in TCAV | 10 minutes
  Percentage of hyper-aerated lung parenchyma defined as lung volume at ≤ - 901 Hounsfield Units (HU) divided by total lung volume, at the end of inspiration in TCAV.
Tidal hyperinflation in TCAV | 10 minutes
  Tidal hyperinflation is defined as the volume of the hyper-aerated (density ≤ - 901 HU) compartment at end-inspiration minus hyper-aerated (density ≤ - 901 HU) volume at end-expiration, and standardized to predicted body weight (PBW), expressed in ml/kg of PBW
Atelectrauma in TCAV and VCV | 10 minutes
  Tidal recruitment of the non-aerated (-100 to +100 Hounsfield Units) compartment was defined as the weight of the non-aerated compartment at end-expiration minus its weight at end-inspiration, and standardized to total lung weight, expressed in %.
Correlation between transpulmonary driving pressure and tidal hyperinflation in TCAV | 10 minutes
  Area under ROC curve of transpulmonary driving pressure to detect cyclic hyperinflation
Correlation between driving pressure and tidal hyperinflation in TCAV | 10 minutes
  Area under ROC curve of driving pressure to detect cyclic hyperinflation

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Pequignot, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU, Nancy, France